CLINICAL TRIAL: NCT03321539
Title: Phase Ⅲ Trial of Concurrent Chemoradiotherapy Followed by Adjuvant Chemotherapy (GP Versus PF) in Patients With N2-3 Nasopharyngeal Carcinoma
Brief Title: Phase Ⅲ Trial of Adjuvant Chemotherapy in Patients With N2-3 Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hai-Qiang Mai,MD,PhD, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-FXY-077
Record Dates: First submitted 2017-07-06; First posted 2017-10-25 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal carcinoma;adjuvant chemotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Intervention Model Description: 1. Cancer Center of Guangzhou Medical University
  2. The Affiliated Hospital of Guizhou Medical University, Guizhou Cancer Hospital
  3. The Affiliated Cancer Hospital of Xiangya School of Medicine, Central South University, Hunan Cancer Hospital
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CCRT+GP (Experimental): Patients receive concurrent cisplatin 100mg/m2 every 21 days for three cycles during radiotherapy followed by adjuvant gemcitabine (1000mg/m2 on day 1 and day 8) and cisplatin (80mg/m2 on day 1) every 21days for three cycles
  Interventions: Drug: CCRT+GP
- CCRT+PF (Active Comparator): Patients receive concurrent cisplatin 100mg/m2 every 21 days for three cycles during radiotherapy followed by adjuvant cisplatin (80mg/m2 on day 1) and 5-fluorouracil (1000mg/m2 civ 96h) every 28 days for three cycles
  Interventions: Drug: CCRT+PF

INTERVENTIONS:
Drug: CCRT+GP — Patients receive concurrent cisplatin 100mg/m2 every 21days for three cycles during Intensity modulated-radiotherapy (IMRT) followed by adjuvant gemcitabine (1000mg/m2 on day 1 and day 8) and cisplatin (80mg/m2 on day 1) every 21 days for three cycles 4 weeks after radiotherapy.
  Other Names: Adjuvant GP
  Arms: CCRT+GP
Drug: CCRT+PF — Patients receive concurrent cisplatin 100mg/m2 every 21 days for three cycles during Intensity modulated-radiotherapy (IMRT) followed by adjuvant cisplatin (80mg/m2 on day 1) and 5-fluorouracil (1000mg/m2 civ 96h) every 28 days for three cycles 4 weeks after radiotherapy.
  Other Names: Adjuvant PF
  Arms: CCRT+PF

SUMMARY:
To see the effect if a combination of concurrent chemoradiotherapy followed by different adjuvant chemotherapy in treating patients with N2-3 nasopharyngeal carcinoma(NPC).

DETAILED DESCRIPTION:
This phase Ⅲ trial is studying how well radiation therapy and chemotherapy work in treating patients with newly diagnosed N2-3 nasopharyngeal cancer. Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as cisplatin and fluorouracil or cisplatin and gemcitabine, work in different ways (concurrent chemoradiotherapy followed by different adjuvant chemotherapy) to stop the growth of tumor cells.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly histologically confirmed non-keratinizing (according to World Health Organization (WHO) histologically type).
* Original clinical staged as any T、N2-3M0（according to the American Joint Committee on Cancer(AJCC) 7th edition）
* No evidence of distant metastasis (M0).
* Age 18-65 years old.
* ECOG Performance status less or equal to 1.
* Adequate marrow: leucocyte count ≥4000/μL, hemoglobin ≥90g/L and platelet count ≥100000/μL.
* Normal liver function test: Alanine Aminotransferase (ALT)、Aspartate Aminotransferase (AST) <1.5×upper limit of normal (ULN) concomitant with alkaline phosphatase (ALP) ≤2.5×ULN, and bilirubin ≤ULN.
* Adequate renal function: creatinine clearance ≥60 ml/min.
* Patients must be informed of the investigational nature of this study and give written informed consent.

Exclusion Criteria:

* WHO Type keratinizing squamous cell carcinoma or basaloid squamous cell carcinoma.
* Age <18 or >65 years.
* Treatment with palliative intent.
* Prior malignancy except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer.
* Pregnancy or lactation.
* History of previous radiotherapy (except for non-melanomatous skin cancers outside intended RT treatment volume).
* Prior chemotherapy or surgery (except diagnostic) to primary tumor or nodes.
* Any severe intercurrent disease, which may bring unacceptable risk or affect the compliance of the trial, for example, unstable cardiac disease requiring treatment, renal disease, chronic hepatitis, diabetes with poor control (fasting plasma glucose >1.5×ULN), and emotional disturbance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2017-10-30 (Actual); Primary Completion 2022-12-25 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Progress-free survival(PFS) | 3 years
  Progress-free survival is calculated from the date of randomization to the date of the first progress at any site or death from any cause or censored at the date of the last follow-up.

SECONDARY OUTCOMES:
Overall survival(OS) | 3 years
  The OS was defined as the duration from the date of random assignment to the date of death from any cause or censored at the date of the last follow-up.
Locoregional failure-free survival(LRRFS) | 3 years
  The LRFS is evaluated and calculated from the date of random assignment until the day of first locoregional relapse or until the date of the last follow-up visit.
Distant metastasis-free survival(DMFS) | 3 years
  The DMFS is evaluated and calculated from the date of random assignment until the day of first distant metastases or until the date of the last follow-up visit.
Overall response rate | 16 weeks after completion of concurrent chemoradiotherapy
  Tumour response was classified according to RECIST, version 1.1
Incidence of acute and late toxicity | 3 years
  Incidence of acute toxicity is calculated for each adverse event respectively and severity is evaluated on basis of Common Terminology Criteria for Adverse Events (CTCAE) 4.0 criteria. Late radiation toxicities were assessed using the Radiation Therapy Oncology Group and European Organization for Research and Treatment of Cancer late radiation morbidity scoring scheme

CONTACTS AND LOCATIONS:
Overall Officials: Hai-Qiang Mai, MD,PhD, Principal Investigator — Sun Yat-sen University
Locations (4):
- China (4):
  - Department of Radiation Oncology, Affiliated Cancer Hospital and Institute of Guangzhou Medical University, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - The Affiliated Hospital of Guizhou Medical University, Guizhou Cancer Hospital, Guiyang, Guizhou
  - The Affiliated Cancer Hospital of Xiangya School of Medicine, Central South University, Hunan Cancer Hospital, Changsha, Hunan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blanchard P, Lee A, Marguet S, Leclercq J, Ng WT, Ma J, Chan AT, Huang PY, Benhamou E, Zhu G, Chua DT, Chen Y, Mai HQ, Kwong DL, Cheah SL, Moon J, Tung Y, Chi KH, Fountzilas G, Zhang L, Hui EP, Lu TX, Bourhis J, Pignon JP; MAC-NPC Collaborative Group. Chemotherapy and radiotherapy in nasopharyngeal carcinoma: an update of the MAC-NPC meta-analysis. Lancet Oncol. 2015 Jun;16(6):645-55. doi: 10.1016/S1470-2045(15)70126-9. Epub 2015 May 6. PMID 25957714
- [Background] Zhang L, Huang Y, Hong S, Yang Y, Yu G, Jia J, Peng P, Wu X, Lin Q, Xi X, Peng J, Xu M, Chen D, Lu X, Wang R, Cao X, Chen X, Lin Z, Xiong J, Lin Q, Xie C, Li Z, Pan J, Li J, Wu S, Lian Y, Yang Q, Zhao C. Gemcitabine plus cisplatin versus fluorouracil plus cisplatin in recurrent or metastatic nasopharyngeal carcinoma: a multicentre, randomised, open-label, phase 3 trial. Lancet. 2016 Oct 15;388(10054):1883-1892. doi: 10.1016/S0140-6736(16)31388-5. Epub 2016 Aug 23. PMID 27567279
- [Background] Chen L, Hu CS, Chen XZ, Hu GQ, Cheng ZB, Sun Y, Li WX, Chen YY, Xie FY, Liang SB, Chen Y, Xu TT, Li B, Long GX, Wang SY, Zheng BM, Guo Y, Sun Y, Mao YP, Tang LL, Chen YM, Liu MZ, Ma J. Concurrent chemoradiotherapy plus adjuvant chemotherapy versus concurrent chemoradiotherapy alone in patients with locoregionally advanced nasopharyngeal carcinoma: a phase 3 multicentre randomised controlled trial. Lancet Oncol. 2012 Feb;13(2):163-71. doi: 10.1016/S1470-2045(11)70320-5. Epub 2011 Dec 7. PMID 22154591
- [Background] Twu CW, Wang WY, Chen CC, Liang KL, Jiang RS, Wu CT, Shih YT, Lin PJ, Liu YC, Lin JC. Metronomic adjuvant chemotherapy improves treatment outcome in nasopharyngeal carcinoma patients with postradiation persistently detectable plasma Epstein-Barr virus deoxyribonucleic acid. Int J Radiat Oncol Biol Phys. 2014 May 1;89(1):21-9. doi: 10.1016/j.ijrobp.2014.01.052. PMID 24725686
- [Result] Ribassin-Majed L, Marguet S, Lee AWM, Ng WT, Ma J, Chan ATC, Huang PY, Zhu G, Chua DTT, Chen Y, Mai HQ, Kwong DLW, Cheah SL, Moon J, Tung Y, Chi KH, Fountzilas G, Bourhis J, Pignon JP, Blanchard P. What Is the Best Treatment of Locally Advanced Nasopharyngeal Carcinoma? An Individual Patient Data Network Meta-Analysis. J Clin Oncol. 2017 Feb 10;35(5):498-505. doi: 10.1200/JCO.2016.67.4119. Epub 2016 Dec 5. PMID 27918720
- [Derived] Liu LT, Liu H, Huang Y, Yang JH, Xie SY, Li YY, Guo SS, Qi B, Li XY, Chen DP, Jin F, Sun XS, Yang ZC, Liu SL, Luo DH, Li JB, Liu Q, Wang P, Guo L, Mo HY, Qiu F, Yang Q, Liang YJ, Jia GD, Wen DX, Yan JJ, Zhao C, Chen QY, Sun R, Tang LQ, Mai HQ. Concurrent chemoradiotherapy followed by adjuvant cisplatin-gemcitabine versus cisplatin-fluorouracil chemotherapy for N2-3 nasopharyngeal carcinoma: a multicentre, open-label, randomised, controlled, phase 3 trial. Lancet Oncol. 2023 Jul;24(7):798-810. doi: 10.1016/S1470-2045(23)00232-2. Epub 2023 Jun 5. PMID 37290468